CLINICAL TRIAL: NCT05859984
Title: A Prospective, Randomized, Double-blind, Double-simulated, Placebo Parallel-controlled, Multicenter Clinical Study on Safety and Efficacy of Recombinant Human Interferon ω Spray in Treatment of Viral Upper Respiratory Tract Infection in Children
Brief Title: To Evaluate the Clinical Efficacy and Safety of Recombinant Human Interferon ω Spray in Treatment of Viral Upper Respiratory Tract Infection in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seventh Medical Center of PLA General Hospital (Other)
Collaborators: The General Hospital of Central Theater Command (Other); The General Hospital of Northern Theater Command (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFNω-VI
Record Dates: First submitted 2023-04-12; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Viral Upper Respiratory Tract Infection
Keywords: Viral Upper Respiratory Tract Infection; recombinant human interferon ω; Safety; Efficacy; 3-12 years

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, double-simulated, placebo parallel-controlled, multicenter design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): 1 bottle of recombinant human interferon ω spray and 1 bottle of placebo（recombinant human interferon ω spray mimics）+base drugs（Xiao'er Changui Tuire granules and Xiao'er Feire Kechuan granules). Each bottle of medication is sprayed once, twice a day. After using the medication, no food or water can be consumed for 20 minutes. Follow the doctor's instructions for use of the base drugs. This treatment course can last up to 7 days.
  Interventions: Drug: recombinant human interferon ω spray
- High dose group (Experimental): 2 bottle of recombinant human interferon ω spray +base drugs（Xiao'er Changui Tuire granules and Xiao'er Feire Kechuan granules). Each bottle of medication is sprayed once, twice a day. After using the medication, no food or water can be consumed for 20 minutes. Follow the doctor's instructions for use of the base drugs. This treatment course can last up to 7 days.
  Interventions: Drug: recombinant human interferon ω spray
- Placebo group (Placebo Comparator): 2 bottle of placebo（recombinant human interferon ω spray mimics）+base drugs（Xiao'er Changui Tuire granules and Xiao'er Feire Kechuan granules). Each bottle of medication is sprayed once, twice a day. After using the medication, no food or water can be consumed for 20 minutes. Follow the doctor's instructions for use of the base drugs. This treatment course can last up to 7 days.
  Interventions: Drug: recombinant human interferon ω spray

INTERVENTIONS:
Drug: recombinant human interferon ω spray — 8 ml/bottle（contain 2 million IU recombinant human interferon ω）

SUMMARY:
To evaluate the clinical efficacy and safety of recombinant human interferon ω spray in treatment of viral upper respiratory tract infection in children aged by 3-12 years, and to explore the appropriate usage and dosage of the drug in treatment of upper respiratory tract infection caused by viruses.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind, double-simulated, placebo parallel-controlled, multi-center clinical study. Children who met the inclusion criteria of viral upper respiratory tract infection in eligible children aged by 3-12 years will be enrolled. The study contained 3 treatment groups. Xiao'er Chaigui Tuire Keli and Xiao'er Feire Kechuan Keli were used as symptomatic treatment drugs in each group, and the two test groups additionally added to different doses of recombinant human interferon ω spray, placebo was added to the placebo group. This study is a prospective, randomized, double-blind, double-simulated, placebo parallel-controlled, multi-center clinical study. Children who met the inclusion criteria of viral upper respiratory tract infection in eligible children aged by 3-12 years will be enrolled. The study contained 3 treatment groups. Xiao'er Chaigui Tuire Keli and Xiao'er Feire Kechuan Keli were used as symptomatic treatment drugs in each group, and the two test groups additionally added to different doses of recombinant human interferon ω spray, placebo was added to the placebo group. In each group, each bottle of drug was sprayed 1 time, sprayed into the child's pharynx, 2 times/dayand should not eat or drink for 20 minutes after using the medicine, Xiao'er Chaigui Tuire Keli and Xiao'er Feire Kechuan Keli should be taken orally according to the doctor's instructions. The treatment period is 7 days. All subjects returned to the study site for evaluating the primary efficacy measures, secondary efficacy measures and safety measures on Treatment Day 7±1. Telephone follow-up was performed on Treatment Day 14±2.

ELIGIBILITY:
Inclusion Criteria:

* 3 years old ≤ age ≤ 12 years old, gender unlimited；
* Routine blood test of white cells < Upper limit of normal value, C reactive protein < Upper limit of normal value. Meeting the description of the diagnostic criteria for viral upper respiratory tract infection in Zhufutang Practical Pediatrics；
* Body temperature ≥ 38 ℃（axillary temperature）；
* The guardian should give informed consent and sign the informed consent form (if the child is ≥ 10 years old, the child should also give informed consent and sign the informed consent form).

Exclusion Criteria:

* Diagnosed as bacterial upper respiratory tract infection.
* Patients with onset time more than 72 hours.
* With severe cardiac, hepatic and renal insufficiency（ALT and AST are 1.5 times above the upper limit of normal value）, abnormal renal function（Scr abnormality） .
* Treated with antiviral drugs orally within two weeks or for external use within one week before inclusion.
* Participated in other clinical trials and took the study medication within one month before inclusion.
* People with low immune function, systemic failure or long-term use of glucocorticoids and immunosuppressants.
* Those who suffer from nervous and mental diseases and cannot cooperate well.
* Allergy constitution（allergic to more than two kinds of drugs or food）or known allergy to interferon and its matrix.
* Because of other diseases that affect the efficacy observer of this study.
* Other conditions considered by the investigator as not appropriate to participate in the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 345 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Complete antipyretic time | 0-7 days post each drug use
  the axillary temperature returns to normal （37.4℃） and remains for 24 h or more.
Incidence of adverse reaction (AR) | 0-14 days post each drug use
  Incidence of adverse reaction (AR)

SECONDARY OUTCOMES:
The effective rate of relieving symptoms of upper respiratory tract infection | 0-7 days post each drug use
  all symptoms of upper respiratory tract infection（nasal congestion, runny nose, sneezing, sore throat, cough）were alleviated efficiently. Judging the severity of the condition through scoring criteria.
Recovery time | 0-7 days post each drug use
  the time required for complete fever relief and all symptoms to be relieved
Use rate of antimicrobial drugs and antipyretic drugs | 0-7 days post each drug use
  Types and frequency of use of antibacterial and antipyretic drugs
Incidence of complications | 0-7 days post each drug use
  Incidence of complications
Recurrence rate of cured subjects | 0-7 days post each drug use
  Recurrence rate of cured subjects
Laboratory examination | 0-7 days post each drug use
  Changes in laboratory indicators，such as red blood cell count; platelet count; glutamic-pyruvic transaminase; urinary protein and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Zhichuan Feng, M.M, Principal Investigator — Seventh Medical Center of PLA General Hospital